CLINICAL TRIAL: NCT05246124
Title: The Effect of Demographic, Mental, and Physical Activity Profiles Towards Burnout in Frontline Healthcare Workers Facing COVID-19 Pandemics in RSUD Dr. Soetomo Surabaya
Brief Title: The Effect of Demographic, Mental, and Physical Activity Profiles Towards Burnout in Frontline Healthcare Workers Facing COVID-19 Pandemics in Dr. Soetomo General Hospital Surabaya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Soetomo General Hospital (Other Government)
Collaborators: Universitas Airlangga (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 0006/KEPK/V/2020
Record Dates: First submitted 2022-02-15; First posted 2022-02-18 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Burnout, Psychological; Anxiety
Keywords: Mental health; COVID-19; Healthcare workers; Anxiety; Burnout; Biomarkers
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders; Psychological Well-Being; COVID-19

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This study used Zumba dance exercise done 3 times a week during 2-week self-isolation period, with each session lasting for 50 minutes. The participants did exercise by following instructions from Zumba video shown
  Interventions: Other: Zumba dance exercise
- Control group (No Intervention): No intervention during 2-week self-isolation period

INTERVENTIONS:
Other: Zumba dance exercise — The intervention was Zumba dance done 3 times a week during the 2-week self-isolation period, with each session lasting for 50 minutes. The participants did exercise by following instructions from Zumba video shown
  Arms: Intervention group

SUMMARY:
This was a randomized controlled trial study to measure the effect of intervention of Zumba dance towards psychological and biological markers in hospital residents managing COVID-19 patients

DETAILED DESCRIPTION:
A study to compare the effect of Zumba dance exercise towards psychological and biological markers in control and intervention groups of residents managing COVID-19 patients. Psychological markers were assessed using State Trait Anxiety Inventory (STAI), Brief Resilience Scale (BRS), and Maslach Burnout Inventory (MBI) questionnaires. Biological markers being measured were neutrophil to lymphocyte ratio (NLR), CD4, Interleukin-6 (IL-6), and salivary cortisol. Measurements were done at the beginning of self-isolation after shift and 2 weeks after self-isolation.

ELIGIBILITY:
Inclusion Criteria:

* Residents of anesthesiology and internal medicine department at Dr. Soetomo General Hospital Surabaya
* Residents managing COVID-19 patients in the special isolation room

Exclusion Criteria:

* Residents that did not fill in the questionnaires completely
* Residents with comorbidities (diabetes, hypertension, heart disease or autoimmune disorders)
* Residents that were infected with COVID-19
* Residents currently or previously diagnosed with psychosis
* Residents refusing to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-06-13 (Actual); Study Completion 2020-06-13 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | 2 weeks
  State anxiety (STAI-S) is the presence subjective feeling of fear and tension, also the occurrence of autonomic nervous activation responding to dangerous or threatening condition. Trait anxiety (STAI-T) is a more stable aspect of tendency towards anxiety, including calmness, self-esteem, and feeling secure. STAI contains 40 statements with the score interpretation ranging from 20-80. The score between 20-37 means having low or no anxiety, 38-44 indicates medium anxiety, and 45-80 suggests high anxiety
Brief Resiliency Scale (BRS) | 2 weeks
  BRS consists of six questions, with three positive statements and three negative statements. Participants choose one of the five responses to the statements, ranging from "strongly disagree" to "strongly agree". There are three categories of results: low
Maslach Burnout Inventory (MBI) | 2 weeks
  The MBI scoring is divided into dimensions of burnout such as emotional exhaustion (EE), depersonalization (DP), and personal accomplishment (PA). The 22-items questionnaire evaluates these domains of burnout, containing 9 items for emotional exhaustion (MBI-EE), 5 items for depersonalization (MBI-DP), and 8 items for personal accomplishment (MBI-PA). Each item is rated using a Likert scale, measuring the experience of the participants, ranging from never (0) to everyday (6). The MBI-EE score consists of high for total score ≥ 30, moderate for 18-28, and low for ≤ 17. The MBI-DP score comprises high for total score ≥ 12, moderate for 6-11, and low for ≤ 5. As for the MBI-PA, it is considered low for a total score ≤ 33, moderate for 34-39, and high for ≥ 40
Cortisol | 2 weeks
  Unstimulated saliva samples, using the passive drooling method, were collected from each participant. The participants should not eat or drink anything at least 1 hour prior to the saliva collection. Also, the participants were instructed to brush their teeth and wash their oral cavities with sterilized water. Samples were kept cold using cooler box and transported to the laboratory. In the laboratory, samples were immediately centrifuged 1700xg at 4°C for 10 minutes within one hour after collection, Samples were aliquoted and stored at -80°C for further analysis of cortisol level.
  Determination of saliva cortisol was performed using a cortisol enzyme immunoassay kit. Samples (25 µL) were treated according to the manufacturer's instructions. The optical density of the samples and standards were measured at a wavelength of 450 nm by a microplate reader
CD4 | 2 weeks
  5 ml blood samples were collected from median cubital vein using a standardized venipuncture technique in EDTA tube for CD4 analysis. Blood samples were centrifuged 2500 rpm for 15 minutes. The serum were then aliquoted and stored at -80°C. CD4 were analyzed by flowcytometry according to the manufacturer's instruction.
Interleukin-6 (IL-6) | 2 weeks
  5 ml blood samples were collected from median cubital vein using a standardized venipuncture technique in serum separator tube (SST) for Interleukin 6. Blood samples were centrifuged 2500 rpm for 15 minutes. The serum were then aliquoted and stored at -80°C. Quantification of Interleukin-6 used commercial ELISA kit according to the manufacturer's instructions. The optical density of the samples and standards were measured by a microplate reader. Samples' concentration was calculated according to the relevant standard curve.
Neutrophil to lymphocyte ratio (NLR) | 2 weeks
  5 ml blood samples were collected from median cubital vein using a standardized venipuncture technique in EDTA tube for NLR analysis. NLR were analyzed by flowcytometry according to the manufacturer's instruction.

CONTACTS AND LOCATIONS:
Overall Officials: Margarita M Maramis, MD, Ph.D, Principal Investigator — Dr. Soetomo General Hospital
Locations (1):
- Dr. Soetomo General Hospital, Surabaya, East Java, Indonesia

IPD SHARING:
Plan to Share IPD: No